CLINICAL TRIAL: NCT03883620
Title: A Phase I, Partially Blind (Observer-blind), Randomized, Single Dose Ascending Study of Dengue Monoclonal Antibody (Dengushield) in Healthy Adults
Brief Title: Safety Study of Dengushield in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Dengushield-01
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Phase 1; Dengue
Keywords: Dengue
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, randomized, partially-blind (observer-blind), placebo controlled, single dose ascending study in healthy adults. For the Cohort 1 (Initial Safety Cohort), no placebo control will be used and hence, blinding is not applicable.
  There will be 4 dose levels. The proposed doses to be studied are; 1 mg/kg, 3 mg/kg, 12 mg/kg and 25 mg/kg. Total of 40 participants will be dosed and followed till Day 84 from dosing.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: For the Cohort 1 (Initial Safety Cohort), no placebo control will be used and hence, blinding is not applicable.For remaining cohorts, both participant and investigator will be unaware of treatment allocation as well as the laboratories analyzing the biochemistry and hematology parameters, pharmacokinetic and immunogenicity (ADA) samples will be blinded to treatment allocation. The drug administrator will be unblinded who will prepare and administer the study drugs. The 7 day safety data for each cohort will be reviewed by group-wise unblinding. Individual level unblinding will be done only in cases of suspected serious adverse reactions as per the judgement of investigator or medical monitor / sponsor representative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Initial Safety Cohort) 1 mg/kg (Experimental): 4 participants will be administered Dengushield at 1 mg/kg body weight as Intravenous injection.
  Interventions: Biological: Dengushield 1 mg/kg (Cohort 1) intravenous
- Cohort 2 Experimental 3mg/kg (Experimental): Initially two participants will be randomized in 1:1 ratio to Dengushield or placebo as a sentinel cohort. If there are no causally related serious safety findings, remaining 10 participants for that cohort will be randomized in 9:1 ratio to Dengushield or placebo.
  Interventions: Biological: Dengushield 3 mg/kg (Cohort 2) intravenous
- Cohort 2 Placebo 3 mg/kg (Placebo Comparator): Initially two participants will be randomized in 1:1 ratio to Dengushield or placebo as a sentinel cohort. If there are no causally related serious safety findings, remaining 10 participants for that cohort will be randomized in 9:1 ratio to Dengushield or placebo and enrolled.
  Interventions: Biological: Placebo 3 mg/kg (Cohort 2) intravenous
- Cohort 3 Experimental 7 mg/kg (Experimental): Initially two participants will be randomized in 1:1 ratio to Dengushield or placebo as a sentinel cohort. If there are no causally related serious safety findings, remaining 10 participants for that cohort will be randomized in 9:1 ratio to Dengushield or placebo.
  Interventions: Biological: Dengushield 7 mg/kg (Cohort 3) intravenous
- Cohort 3 Placebo 7 mg/kg (Placebo Comparator): Initially two participants will be randomized in 1:1 ratio to Dengushield or placebo as a sentinel cohort. If there are no causally related serious safety findings, remaining 10 participants for that cohort will be randomized in 9:1 ratio to Dengushield or placebo.
  Interventions: Biological: Placebo 7 mg/kg (Cohort 3) intravenous
- Cohort 4 Experimental 12 mg/kg (Experimental): Initially two participants will be randomized in 1:1 ratio to Dengushield or placebo as a sentinel cohort. If there are no causally related serious safety findings, remaining 10 participants for that cohort will be randomized in 9:1 ratio to Dengushield or placebo.
  Interventions: Biological: Dengushield 12 mg/kg (Cohort 4) intravenous
- Cohort 4 Placebo 12 mg/kg (Placebo Comparator): Initially two participants will be randomized in 1:1 ratio to Dengushield or placebo as a sentinel cohort. If there are no causally related serious safety findings, remaining 10 participants for that cohort will be randomized in 9:1 ratio to Dengushield or placebo.
  Interventions: Biological: Placebo 12 mg/kg (Cohort 4) intravenous

INTERVENTIONS:
Biological: Dengushield 1 mg/kg (Cohort 1) intravenous — Participants will be administered Dengushield 1 mg/kg as slow intravenous injection.
  Arms: Cohort 1 (Initial Safety Cohort) 1 mg/kg
Biological: Dengushield 3 mg/kg (Cohort 2) intravenous — Participants will be administered Dengushield 3 mg/kg as slow intravenous infusion.
  Arms: Cohort 2 Experimental 3mg/kg
Biological: Placebo 3 mg/kg (Cohort 2) intravenous — Participants will be administered Placebo 3 mg/kg as slow intravenous infusion.
  Arms: Cohort 2 Placebo 3 mg/kg
Biological: Dengushield 7 mg/kg (Cohort 3) intravenous — Participants will be administered Dengushield 7 mg/kg as slow intravenous infusion.
  Arms: Cohort 3 Experimental 7 mg/kg
Biological: Placebo 7 mg/kg (Cohort 3) intravenous — Participants will be administered Placebo 7 mg/kg as slow intravenous infusion.
  Arms: Cohort 3 Placebo 7 mg/kg
Biological: Dengushield 12 mg/kg (Cohort 4) intravenous — Participants will be administered Dengushield 12 mg/kg as slow intravenous infusion.
  Arms: Cohort 4 Experimental 12 mg/kg
Biological: Placebo 12 mg/kg (Cohort 4) intravenous — Participants will be administered Placebo 12 mg/kg as slow intravenous infusion.
  Arms: Cohort 4 Placebo 12 mg/kg

SUMMARY:
This Phase 1 study to evaluate the safety of a single dose of Dengushield (dengue monoclonal antibody) in healthy adults.

DETAILED DESCRIPTION:
This Phase 1 study will evaluate the safety and tolerability of a single dose of Dengushield (dengue monoclonal antibody) in healthy adults in a dose-escalating study design. In addition, pharmacokinetics will also be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18-45 years, men, or women.
2. Negative Dengue NS1 at screening indicating no current dengue infection
3. Seronegative for dengue IgG
4. Participants who are willing to comply with the requirements of the study protocol and attend scheduled visit.
5. Participants who give written informed consent.
6. Participants having laboratory parameters within normal range
7. Participants with Body Mass Index (BMI) between 18 to 30 (both inclusive)
8. Satisfactory baseline medical assessment as assessed by physical examination and normal laboratory values or minor variations that is acceptable for study entry.

Exclusion Criteria:

1. Presence of acute infection in the preceding 14 days or presence of a temperature ≥ 38.0°C, or acute symptoms of infection greater than of "mild" severity on the scheduled date of first dosing
2. History or presence of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, autoimmune, dermatologic or immunosuppressive disorders.
3. Evidence of any other significant active haematological disease, or having donated > 450 mL of blood within the past three months.
4. Evidence or history of substance abuse including alcohol, or previous substance abuse within the last year.
5. Participation or planned participation in a study involving the administration of an investigational compound within the past one month or during this study period.
6. Planned administration of any vaccine not foreseen by the study protocol 4 weeks before and after dosing except for influenza vaccination.
7. Receipt of immunoglobulins and/or any blood products within 9 months of study enrolment or planned administration of any of these products during the study period.
8. Laboratory confirmed infection with hepatitis B virus (HBsAg positive), hepatitis C virus (anti-HCV positive) or human immunodeficiency virus (HIV positive) at screening.
9. History of allergic disease, allergic reactions or known hypersensitivity to any component of the study product (Mild non-medication allergies allowed).
10. Known bleeding disorders.
11. Women who are pregnant, breast-feeding, or considering becoming pregnant.
12. Any condition that, in the opinion of the investigator, would complicate or compromise the study or well-being of the participant.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with post-injection/ infusion adverse events (AEs) including hypersensitivity reaction, anaphylactic reaction and other AEs occurring within 4 hours of the start of dosing | 4 hours post administration of drug
  Safety monitoring for 4 hours
The proportion of participants with AEs, discontinuations due to AEs, and serious adverse events (SAEs) | 84 days
  Safety
Proportion of participants with clinically significant abnormal safety laboratory (hematology and chemistry parameters) findings | 28 days
  Safety

SECONDARY OUTCOMES:
Time to maximum serum concentration of Dengushield - Tmax | 84 days
  Time to maximum serum concentration of Dengushield - Tmax
Presence or absence of anti-Dengushield antibody in sera samples | 84 days
  Anti-Dengushield antibodies will be checked in sera samples.
Maximum serum concentration of dengushield - Cmax | 84 days
  Maximum serum concentration of dengushield
AUC from time 0 to infinity of Dengushield | 84 days
  Area under curve of Dengushield from time 0 to infinity (AUC0-infinity)
AUC from time 0 to 84 days of Dengushield | 84 days
  Area under curve of Dengushield from time 0 to 84 days (AUC0-84d)
Half life of Dengushield - t1/2 | 84 days
  Half life of Dengushield
Volume of distribution of Dengushield | 84 days
  Volume of distribution of Dengushield
Clearance of dengushield | 84 days
  Clearance of dengushield
Elimination rate constant of dengushield | 84 days
  Elimination rate constant of dengushield

CONTACTS AND LOCATIONS:
Overall Officials: Prasad Kulkarni, MD, Study Director — Serum Institute of India Pvt. Ltd.
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gunale B, Farinola N, Kamat CD, Poonawalla CS, Pisal SS, Dhere RM, Miller C, Kulkarni PS. An observer-blind, randomised, placebo-controlled, phase 1, single ascending dose study of dengue monoclonal antibody in healthy adults in Australia. Lancet Infect Dis. 2024 Jun;24(6):639-649. doi: 10.1016/S1473-3099(24)00030-6. Epub 2024 Feb 23. PMID 38408457